CLINICAL TRIAL: NCT05134623
Title: Smurf2 Gene Expression in Urinary Tract Tumors - Tissue Immunohistochemitry and Urinary Sediment Analysis
Brief Title: Smurf2 Gene Expression in Urinary Tract Tumors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Collaborators: Azrieli Faculty of medicine, Bar Ilan University, Safed, IL (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0029-20-ZIV
Record Dates: First submitted 2021-11-14; First posted 2021-11-26 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Bladder Neoplasm
Keywords: bllader neoplasm,; SMURF2; biomarker; urinary sediment; immunohistochemistry; PCR
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — parafin sections of bladder tumors obtained during trans urethral resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: immunohistochemistry of tumors samples — routine resection of tumors, further analysis and immunohisochemical staining of the tissue slides.

SUMMARY:
Smurf2 and bladder cancer - research proposal summary The Smurf2 gene was recently identified as a tumor suppressor gene. It is an E3 ubiquitin ligase and carries a significant role in major cellular processes such as cell division, genomic stability, DNA repair as well as resistance to anti-tumoral drugs.

Recent studies showed that in several common tumors (prostate, breast, osteosarcoma etc.), a significant decrease in the expression or activity of Smurf2 can be noted, making the cells more susceptible to malignant transformation and the tumors more aggressive and highly resistant to various medications.

Bladder cancer is no. 4 cancer in men and 6 in women, and a major cause of cancer related death. Common risk factors are smoking and occupational exposure to aniline dyes or aromatic amines. Its' most common presentation is painless hematuria. Once the diagnosis of a bladder tumor is made, endoscopic resection of the tumors is performed. Superficial tumors of low malignancy may be treated by repeated resections, highly malignant tumors require additional therapy and aggressive tumors invading the bladder muscle layer require radical surgery and chemo-radiotherapy. Therefore, all patients are closely monitored by repeated cystoscopies (endoscopic inspection of the bladder), each 3 months, lifelong.

In an effort to minimize patients' discomfort, there is a constant search for a reliable biomarker in the urine of patients. A marker with good sensitivity and specificity will predict in a noninvasive fashion early recurrence or absence of bladder tumors, sparing the need for invasive cystoscopy. The presence of a biomarker may be used as prognostic factor or a measure of response to therapy.

The aim of this research is to characterize the presence of smurf2 in bladder tumors and determine whether it may be utilized as a reliable biomarker for bladder cancer.

DETAILED DESCRIPTION:
Smurf2 and bladder cancer - research proposal summary - detailed

The Smurf2 gene was recently identified as a tumor suppressor gene. It is an E3 ubiquitin ligase and carries a significant role in major cellular processes such as cell division, genomic stability, DNA repair as well as resistance to anti-tumoral drugs.

Recent studies showed that in several common tumors (prostate, breast, osteosarcoma etc.), a significant decrease in the expression or activity of Smurf2 can be noted, making the cells more susceptible to malignant transformation and the tumors more aggressive and highly resistant to various medications.

Bladder cancer is no. 4 cancer in men and 6 in women, and a major cause of cancer related death. Common risk factors are cigarrete smoking and occupational exposure to aniline dyes or aromatic amines. Its' most common presentation is painless hematuria. Once the diagnosis of a bladder tumor is made, endoscopic resection of the tumors is performed. Superficial tumors of low malignancy may be treated by repeated resections, highly malignant tumors require additional therapy and aggressive tumors invading the bladder muscle layer require radical surgery and chemo-radiotherapy. Therefore, all patients are closely monitored by repeated cystoscopies (endoscopic inspection of the bladder.

In an effort to minimize patients' discomfort, there is a constant search for a reliable biomarker in the urine of patients. A marker with good sensitivity and specificity will predict in a noninvasive fashion early recurrence or absence of bladder tumors, sparing the need for invasive cystoscopy. The presence of a biomarker may be used as prognostic factor or a measure of response to therapy.

The aim of this research is to characterize the presence of smurf2 in bladder tumors and determine whether it may be utilized as a reliable biomarker for bladder cancer.

In the study, the investigators will collect samples from bladder tumors of patient referred for transurethral resection of a known bladder tumor. The tissue will be processed routinely yet additional slides will be performed and used for immunohistochemical analysis. The investigators will characterize the expression of SMURF2 in the tissue, its abundance, the distribution between the nucleus and cytoplasm and possible differences between the tumors tissue and surrounding normal margins.

Further on, the investigators will collect urine samples from patients with these tumors and examine the urinary sediment using PCR and proteomic examination. The data will be used for further research using the SMURF2 product as a possible novel bio-marker for the presence of bladder tumors and for non-invasive detection and follow-up of patients on surveillance following surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Identified bladder tumor
* Scheduled for transurethral resection
* Informed consent

Exclusion Criteria:

* Previous bladder, prostate or pelvic irradiation
* Persistent urinary tract infection
* Intravesical therpy with BCG within 6 months prior to surgery.
* Intravesical chemotherapy within 6 months prior to surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients, diagnosed with bladder tumors, referred for transurethral resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Smurf2 and bladder cancer | 6 months
  The presence of SMURF2 in bladder tumor tissue compared to normal surrounding tissue

SECONDARY OUTCOMES:
Smurf2 and bladder cancer | 6 months
  The distribution of SMURF2 in bladder tumor cells - nucleus to cytoplasm
Smurf2 and bladder cancer | 6 months
  Identification of the SMURF2 product in the urinary sediment using proteomics and PCR

CONTACTS AND LOCATIONS:
Overall Officials: Ran Katz, MD, Study Director — Ziv Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manikoth Ayyathan D, Koganti P, Marcu-Malina V, Litmanovitch T, Trakhtenbrot L, Emanuelli A, Apel-Sarid L, Blank M. SMURF2 prevents detrimental changes to chromatin, protecting human dermal fibroblasts from chromosomal instability and tumorigenesis. Oncogene. 2020 Apr;39(16):3396-3410. doi: 10.1038/s41388-020-1226-3. Epub 2020 Feb 26. PMID 32103168